CLINICAL TRIAL: NCT05676060
Title: X-ray Guided Facet Block in Chronic Low Back Pain
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nada Tarek, Dr, Assiut University
Other Study IDs: Facet block
Record Dates: First submitted 2022-12-22; First posted 2023-01-09 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2022-12

CONDITIONS: Back Pain
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

INTERVENTIONS:
Combination Product: quasi — block facet joint in back pain due to afacet cause
  Other Names: facet block

SUMMARY:
Review outcome of injection of facet joint in chronic low back pain

DETAILED DESCRIPTION:
Low back pain is a common problem that most people may experience. the incidence of low back pain is highest in the third decade and increases with age until the 60-65 year age group.

In the USA the prevalence of Low back pain is between 15 and 45%. Facet joint is the primary cause of pain in 10-15% of young adult patients with chronic low back pain.

Probable risk factors include genetic factors, age, smoking, heavy physical work, static work postures, lifting, vibration, obesity, and psychosocial factors.(2) Other Causes of low back pain include muscle and ligament strain, bulging or ruptured disc, arthritis, osteoporosis Treatment of chronic low back pain include pharmacological treatment, ,epidural steroid injection ,facet joint block and back surgery The facet joints are a set of plane types of synovial joints between the articular processes of two adjacent vertebrae, The lumbar facet joint is innervated by the medial branch from the posterior ramus of the lumbar spinal nerve.

Lumbar facet joint injections are performed by various techniques, including fluoroscopic-guided technique indications of diagnostic and therapeutic facet joint interventions

1. Average pain levels > 5 on a scale of 0 to 10.
2. Contraindications or inability to undergo physical therapy or inability to tolerate oral medications.

Complications from facet joint injections in the lumbar spine are rare and mostly related to the needle placement and/or reactions to injected drugs.(3)

ELIGIBILITY:
Inclusion criteria:1-strong clinical suspicion of the facet syndrome,

2-Focal tenderness over the facet joints

3-Low back pain with normal radiological findings,

4-Post-laminectomy syndrome with no evidence of arachnoiditis or recurrent disc disease,

5-Persistent low back pain after lumbar spinal 6- Failed conservative treatment, including physical therapy with exercises, chiropractic management, and pharmacologic therapy

Exclusion Criteria:

- 1- Low back pain with abnormal radiological findings,

2-Post-laminectomy syndrome with evidence of arachnoiditis or recurrent disc disease,

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: individual
Sampling Method: Probability Sample
Enrollment: 43 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale | Baseline
  The pain VAS is a unidimensional measure of pain intensity, used to record patients' pain progression, or compare pain severity between paints with similar conditions. VAS has been widely used in diverse adult populations